CLINICAL TRIAL: NCT02618317
Title: Comparison of Effectiveness and Safety of Three Lock Solutions for Long-Term Central Venous Catheter for Hemodialysis
Acronym: CLOCK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marcus Vinicius de Souza Joao Luiz, MSc., Pharm.D., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USaoPaulo CLOCK
Record Dates: First submitted 2015-09-18; First posted 2015-12-01 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Kidney Disease
Keywords: renal dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Heparin Lock Solution (Active Comparator): Patients on Heparin 1,000 U/ml locking solution, administered at the end of each dialysis session during a 15-week period .
  Interventions: Drug: Heparin Lock Solution
- Trissodium Citrate 30% (Experimental): Patients on trissodium citrate 30% locking solution, administered at the end of each dialysis session during a 15-week period .
  Interventions: Drug: Trissodium Citrate 30%
- Minocycline-EDTA 30 mg/ml - 3 mg/ml (Experimental): Patients on Minocycline 30 mg/ml/EDTA 3 mg/ml locking solution, administered at the end of each dialysis session during a 15-week period.
  Interventions: Drug: Minocycline-EDTA 30 mg/ml - 3 mg/ml

INTERVENTIONS:
Drug: Heparin Lock Solution — Just after the insertion (since first the hemodialysis session), long-term Central Venous Catheter of CKD 5D patients on high-efficiency hemodialysis have been locked during 15 weeks (100 days) with appropriate lock solution.
  Other Names: Hemofol (Traade Mark)
  Arms: Heparin Lock Solution
Drug: Trissodium Citrate 30% — ust after the insertion (since first the hemodialysis session), long-term Central Venous Catheter of CKD 5D patients on high-efficiency hemodialysis have been locked during 15 weeks (100 days) with appropriate lock solution.
  Other Names: CitraLock(Trade Mark)
  Arms: Trissodium Citrate 30%
Drug: Minocycline-EDTA 30 mg/ml - 3 mg/ml — ust after the insertion (since first the hemodialysis session), long-term Central Venous Catheter of CKD 5D patients on high-efficiency hemodialysis have been locked during 15 weeks (100 days) with appropriate lock solution.
  Other Names: Cath-Safe (Trade Mark)
  Arms: Minocycline-EDTA 30 mg/ml - 3 mg/ml

SUMMARY:
Background: Poor flow (PF) and catheter-related blood stream infections (CRBSI) are highly prevalent among CKD 5D patients with long-term central venous catheters. Heparin (H) catheter lock solutions are commonly used to maintain catheter patency, however PF and CRBSI incidence remains high. The purpose of this study was to evaluate two lock solutions on reduction of PF and CRBSI: one, a lock solution combining of the tetracycline antibiotic minocycline with the anticoagulant/chelation agent EDTA (M-EDTA) versus H; and other, trisodium citrate (C) versus H. M-EDTA and C were also evaluated as to their safety versus H.

Methods:As regards the pilot project, thirty CKD 5D patients on high-efficiency hemodialysis (blood flow rate = 350 ml/min) at the Integrated Centre of Nephrology (Guarulhos, Brazil) were randomized 1:1:1 to receive M-EDTA, C or H locks for 15 weeks. Lock solutions concentrations were M-EDTA 30 mg/ml/3 mg/ml, C 30% (C) and H 1,000 U/ml and both investigators and patients were blinded to treatment allocation. The primary end-point was a 10% reduction in HD blood flow rates (35ml). The frequency of CRBSI was recorded. Bleeding and lock solution-related adverse events were the primary safety end points. Logistic Regression was performed to evaluate differences in PF rates among the treatments (SPSS version 13.0, IBM, USA).

Based upon the pilot-study data, the clinical trials has being executed in order to verify whether the three lock solutions have the same performance or not.

DETAILED DESCRIPTION:
Methods: 75 CKD 5D patients on high-efficiency hemodialysis (blood flow rate = 350 ml/min) at the Integrated Centre of Nephrology (Guarulhos, Brazil) will be randomized 1:1:1 to receive M-EDTA, C or H locks for 15 weeks. Lock solutions concentrations are M-EDTA 30 mg/ml/3 mg/ml, C 30% (C) and H 1,000 U/ml and both investigators and patients are blinded to treatment allocation. The primary end-point is a 10% reduction in HD blood flow rates (35ml). The frequency of CRBSI will be recorded. Poor Flow Rate (event/1,000 catheter-day) and CRBSI Rate (event/1,000 catheter-day) will be calculated in each arm. Bleeding and lock solution-related adverse events are also the primary safety end points and their rates (events/1,000 catheter-day) will be calculated. Logistic Regression will be performed to evaluate differences in PF, CRBSI, Bleeding and lock solution-related adverse events rates among the treatments (SPSS version 13.0, IBM, USA).

ELIGIBILITY:
Inclusion Criteria:

* male and female patients;
* patients with subclavian long term central venous catheter;
* patients on on high-efficiency hemodialysis (BFR= 350 ml; dialisate flow = 500 ml; 3 times; 4-hour sessions).

Exclusion Criteria:

* pregnant; patients on oral coagulants; patients aged less than 18 years;
* patients aged more than 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Poor Blood Flow Rate(BFR) | 100 days
  Reduction of 35 ml in the BFR of 2350 ml on hemodialysis is considered a primary endpoint for this trial

SECONDARY OUTCOMES:
Adverse Drug Reactions Related to lock solutions (ADR) | 100 days
  ADR is considered secondary endpoint for this trial
Cather-Related Blood Stream Infection (CRBSI) | 100 days
  CRBSI is considered secondary endpoint for this trials

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Luiz, MSc, PharmD, Principal Investigator — PhD student
Locations (1):
- Integrated Centre of Nephrology, Guarulhos, São Paulo, Brazil